CLINICAL TRIAL: NCT05927233
Title: Effect of Methylprednisolone on Systemic Inflammatory Response and Clinical Parameters During Pediatric Congenital Open-Heart Surgery: A Randomized Controlled Trial
Brief Title: Effect of Methylprednisolone on Systemic Inflammatory Response During Pediatric Congenital Open-Heart Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Saad Yousuf, Senior Instructor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-6247-18639
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cyanotic Heart Disease; Cardiopulmonary Bypass
Keywords: Paediatric population
MeSH Terms: interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Experimental): IV Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Group P (Placebo Comparator): IV Normal Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Methylprednisolone — 30 ml Methylprednisolone (30mg/kg) with a maximum dose of 500 mg
  Arms: Group M
Drug: Saline — 30 ml Normal saline
  Arms: Group P

SUMMARY:
The goal of this study is to evaluate the effects of steroids on the early postoperative inflammatory response in patients undergoing elective pediatric congenital cardiac surgery, requiring cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* Children 1 month- 18 years of age
* Undergoing Cardiac surgery for the first time and requiring CPB
* Surgeries for both cyatonic and acyanotic heart disease

Exclusion Criteria:

* Pre-mature babies (< 28 weeks at birth)
* Neonates
* Prior cardiac requiring CPB
* Surgeries requiring CPB > 6 hours
* Surgeries requiring second run of CPB
* Patients requiring additional steroids during first 24 hours of CICU stay
* Patient expires within the initial 24 hours CICU stay.
* Compromised immune system - that is, known immunodeficiency or use of
* immunomodulatory therapy.
* Peri-operative presence of two or more clinical or laboratory signs of active infection that were not attributable to any other cause: fever more than 100°F, heart rate or respiratory rate more than the normal range for age, white blood cell count more than 15% of the upper limit of normal, and an elevated C-reactive protein level above baseline.
* Preoperative mechanical ventilation, and preoperative need of inotropic agents or mechanical circulatory support.
* Patient already receiving steroids

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum levels of Interleukin- 6 | Before the first dose of steroid), second sample will be drawn after immediately protamine infusion, third sample at 24 hours after CPB and the fourth sample will be drawn at 48 hours after CPB
  serum levels of Interleukin- 6 will be measured using ELISA
Serum levels of CRP | Before the first dose of steroid), second sample will be drawn after immediately protamine infusion, third sample at 24 hours after CPB and the fourth sample will be drawn at 48 hours after CPB
  serum levels of CRP will be measured using ELISA

SECONDARY OUTCOMES:
Serum creatinine level | Before the first dose of steroid), second sample will be drawn after immediately protamine infusion, third sample at 24 hours after CPB and the fourth sample will be drawn at 48 hours after CPB

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keski-Nisula J, Pesonen E, Olkkola KT, Peltola K, Neuvonen PJ, Tuominen N, Sairanen H, Andersson S, Suominen PK. Methylprednisolone in neonatal cardiac surgery: reduced inflammation without improved clinical outcome. Ann Thorac Surg. 2013 Jun;95(6):2126-32. doi: 10.1016/j.athoracsur.2013.02.013. Epub 2013 Apr 18. PMID 23602068
- [Background] Gibbison B, Villalobos Lizardi JC, Aviles Martinez KI, Fudulu DP, Medina Andrade MA, Perez-Gaxiola G, Schadenberg AW, Stoica SC, Lightman SL, Angelini GD, Reeves BC. Prophylactic corticosteroids for paediatric heart surgery with cardiopulmonary bypass. Cochrane Database Syst Rev. 2020 Oct 12;10(10):CD013101. doi: 10.1002/14651858.CD013101.pub2. PMID 33045104